CLINICAL TRIAL: NCT06125093
Title: Early Treatment for Children With Mental Health Problems and Genetic Abnormalities Through a Parenting Intervention (The GAP): A Pragmatic Randomized Controlled Trial
Brief Title: Study of an Early Parenting Intervention for Children With Genetic Abnormalities and Mental Health Problems
Acronym: The GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other); Parc Taulí Hospital Universitari (Other); Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-168-22; 434/U/2022 (Other Grant/Funding Number: Fundació La MaratóTV3)
Record Dates: First submitted 2023-10-23; First posted 2023-11-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Genetic Syndrome; Language Development; Autism or Autistic Traits; Parenting
Keywords: early intervention; parenting; randomized controlled trial; pragmatic; genetic syndromes; mental health; development
MeSH Terms: conditions — Genetic Diseases, Inborn; Autistic Disorder; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Those in the intervention group will participate in a weekly group-based online intervention for approximately 6 months (Incredible Years-Autism Spectrum and Language Delays Parent Program, IY-ASLD®).
  Families allocated to the intervention group will also receive treatment as usual (TAU).
  Interventions: Behavioral: Incredible Years Autism Spectrum and Language Delays Parent Program (IY-ASLD®)
- Treatment as usual (TAU) group (No Intervention): The TAU condition involves outpatient appointments with different paediatric specialists in the hospitals of the 3 sites of the study.
  Depending on the patients' needs, some cases will be assisted in early years centers or child mental health centers based in the community.

INTERVENTIONS:
Behavioral: Incredible Years Autism Spectrum and Language Delays Parent Program (IY-ASLD®) — The IY-ASLD® program is a weekly group-based intervention for parents of children presenting neurodevelopmental problems (ASD symptoms, communication or language difficulties). The group is formed by 6-10 parents, and it is led by a group leader and a co-therapist, trained in the model.
  The intervention is manualized. It includes video modelling and emphasizes the importance of practice-based learning through role-playing. The IY-ASLD® program takes into consideration the different developmental levels of each child and pairs parents according to this variable in role-play and other one-to-one discussions. Weekly home tasks will be assigned to parents, and families will be phoned each week to encourage home-based practice.
  The intervention will be conducted online. Even though the IY-ASLD® original intervention comprises 14 sessions, the online format requires 22 weekly sessions.
  Fidelity to the intervention will be assessed in accordance with the regulations of the program.
  Other Names: Parenting intervention
  Arms: Intervention group

SUMMARY:
The GAP study is a randomized controlled trial that aims to determine the feasibility and efficacy of the "Incredible Years Autism Spectrum and Language Delays" (IY-ASLD®) intervention for families of children with developmental problems from a genetic basis. It is a multicentric trial where families will randomly be assigned to the intervention group or to a control group (they will follow their usual treatment). The intervention will be carried out in an online format, and it will involve 22 weekly group sessions. The results of The GAP study will help clinicians and policy makers in guiding towards evidence-based treatment options for these particularly vulnerable group of infants.

DETAILED DESCRIPTION:
Children born with genetic abnormalities have higher risk of presenting developmental and mental health problems. Their parents tend to express higher anxiety levels, as parenting children with developmental problems can be a stressful challenge for many families. These infants can present important behaviour, emotion regulation and social interaction problems. These problems usually have a complex clinical presentation determined by their genetic abnormality. Despite many of their impairing symptoms can overlap with the characteristics of the Autism Spectrum Disorder (ASD), in many cases they do not meet criteria for a full-blown ASD diagnosis. These patients are placed in a double disadvantaged situation, as on top of suffering a genetic disease, they do not usually enter the ASD care-pathways and do not have access to effective therapies for their impairing symptoms. This problem should be addressed, as there is wide scientific evidence on early parenting programs that improve infants' developmental problems and parents' mental health. These parenting programs are structured interventions that provide parenting skills to improve the acquisition of children's social and emotion regulation abilities. Such interventions have been widely implemented internationally, but unfortunately, most families treated within our mental health system still do not have access to them. A good example is the parenting program "Incredible Years Autism Spectrum and Language Delays (IY-ASLD®)", focused on improving young children's development and parental stress levels. Recently, the feasibility and acceptability of implementing this program in different areas of the national territory has been studied, with high satisfaction levels expressed by participant families (parents of children with language delays or ASD). However, the scientific evidence is very limited for children with developmental problems from a genetic basis, particularly for those with dysfunctional symptoms' that do not meet diagnostic threshold for an ASD diagnosis.

The GAP study aims to determine, for the first time, the feasibility and efficacy of the IY-ASLD® intervention for families of children with developmental problems from a genetic basis. It is a multicentric randomized controlled trial where families will randomly be assigned to the intervention group or to a control group (they will follow their usual treatment). As genetic abnormalities are rare, clinicians will carry out the intervention in an online format (22 weekly sessions), reaching out all affected families that live scattered throughout the national territory. The results of The GAP study will help clinicians and policy makers in guiding towards evidence-based treatment options for these particularly vulnerable group of infants.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3.0 - 7.11 years at recruitment
2. Children with a diagnosis or in diagnostic process for high suspicion of a genetic abnormality
3. For children up to 5.11 years with withdrawn (defined as CBCL/1.5-5 scores above the borderline clinical range, T-score> 65) AND/OR pervasive developmental problems (defined as CBCL/1.5-5 scores above the borderline clinical range, T-score> 65) AND/OR socialization difficulties (defined as Vineland-III scores below 1SD in the socialization subdomains).
4. For children over 6 years with social problems (defined as CBCL/6-18 scores above the borderline clinical range, T-score> 65) AND/OR thought problems (defined as CBCL/6-18 scores above the borderline clinical range, T-score> 65) AND/OR socialization difficulties (defined as Vineland-III scores below 1SD in the socialization subdomains).
5. Parents/caregivers showing good understanding of the Spanish or Catalan language
6. Parents/caregivers consenting to take part in the study and signing the informed consent

Exclusion Criteria:

1. Children diagnosed with an Autism Spectrum Disorder
2. Children scoring above diagnostic cut-off for Autism or Autism Spectrum Disorder in the ADOS-2.
3. Attending another structured parenting program
4. Children in the care of their local authority

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Percentage of parents engaging with and finishing the program | Attendance sheet completed weekly throughout treatment (22 weeks total)
  Parents' attendance at the sessions will be regeristered weekly with a sheet of attendance, with the aim to determine levels of compliance and engagement with the intervention. An attendance of at least 15/22 sessions is expected, with a minimum of 50% of parents finishing the program.
Compliance and satisfaction throughout the study (Autism Program Parent Weekly Evaluation) | Questionnaire administered to the intervention group weekly throughout treatment (22 weeks total)
  Parents' compliance and satisfaction with the intervention will be assessed weekly after each session with the questionnaire "Autism Program Parent Weekly Evaluation", which is part of the IY-ASLD® program materials.
Parents' acceptability and satisfaction with the program (evaluated with the Autism Program Parent Final Satisfaction Questionnaire) | Administered to the intervention group at treatment completion (approximately 22 weeks after baseline)
  Parents' acceptability and satisfaction with the program will be assessed with the Autism Program Parent Final Satisfaction Questionnaire (included within the IY-ASLD® program). Data will be collected after the last session of the intervention.
Parents' overall experiences with the program (evaluated with individual interviews) | Interviews to the participants of the intervention group at treatment completion (approximately 22 weeks after baseline)
  Individual interviews will be conducted after the last session of the intervention to explore from a qualitative perspective: (1) parents' acceptability, satisfaction and overall experience with the intervention, and (2) parents' perceived changes in their parenting skills and parental distress after the intervention.
  Outcome measurements 3 and 4 will be combined to determine parents' experiences, acceptability and satisfaction with the program.

SECONDARY OUTCOMES:
Changes from baseline to post-intervention in Parent Stress Inventory-Short Form (PSI-SF) | Administered to the intervention and control group at baseline (prior to programme initiation) and at immediately after the intervention (approximately 22 weeks after baseline)
  The PSI-SF is a 36-item questionnaire that specifically focuses on assessing parental stress associated with the care of their offspring. It has three domains: parental distress, parent-child dysfunctional interaction, and difficult child, which combine to form a total stress scale. This tool will be administered before and after the intervention. It has shown good internal consistency.
Changes from baseline to post-intervention in Alabama Parenting Questionnaire-Preschool revision (APQ-Pr) | Administered to the intervention and control group at baseline (prior to programme initiation) and at immediately after the intervention (approximately 22 weeks after baseline)
  The APQ-Pr is a 32-item parent-reported questionnaire measuring parenting practices that are consistently associated with disruptive child behaviors. This version has 3 dimensions: positive parenting, inconsistent parenting, and punitive parenting. It will be collected before and after the intervention. This measure has shown good internal consistency and validity.
Changes from baseline to post-intervention in Beck Depression Inventory (BDI) | Administered to the intervention and control group at baseline (prior to programme initiation) and at immediately after the intervention (approximately 22 weeks after baseline)
  The BDI is a 21-item screening tool assessing the severity of depressive symptoms. It is a standardized and validated questionnaire, often used in mood disorder assessments. It will be collected before and after the intervention. It has good reliability.
Changes from baseline to post-intervention in Autism-Specific Five Minute Speech Sample (ASFMFSS) | Administered to the intervention and control group at baseline (prior to programme initiation) and at immediately after the intervention (approximately 22 weeks after baseline)
  ASFMFSS is a narrative 5-min interview used to measure parental-expressed emotions for children with ASD and related disorders. Parents are asked to speak about their child and the parent-child relationship. Speech samples are audiotaped, transcribed, and coded following four global categories: (a) initial statement, (b) warmth, (c) relationship, (d) emotional over-involvement, (e) critical comments, and (f) positive comments. Expressed emotions will be measured before and after the intervention. Inter-rater reliability and code-recode reliability of this measure have been shown to be good to excellent.
Clinicians' experiences with the intervention delivered | Interviews to clinicians at treatment completion (approximately 22 weeks after baseline)
  Individual interviews will be conducted after the last session with clinicians who delivered the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laia Villalta, MD, PhD, Principal Investigator — Hospital Sant Joan de Déu. Fundació Privada per a la Recerca i la Docència Sant Joan de Déu; Anna Maria Cueto-González, MD, Study Chair — Hospital Universitari Vall d'Hebron. Vall d'Hebron Institut de Recerca; Carmen Manso, MD, Study Chair — Parc Taulí Hospital Universitari; Mercedes Serrano, MD, PhD, Study Chair — Hospital Sant Joan de Deu
Locations (3):
- Spain (3):
  - Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valencia F, Urbiola E, Romero-Gonzalez M, Navas I, Elias M, Garriz A, Ramirez A, Villalta L. Protocol for a randomized pilot study (FIRST STEPS): implementation of the Incredible Years-ASLD(R) program in Spanish children with autism and preterm children with communication and/or socialization difficulties. Trials. 2021 Apr 20;22(1):291. doi: 10.1186/s13063-021-05229-1. PMID 33879224
- [Background] Landa RJ. Efficacy of early interventions for infants and young children with, and at risk for, autism spectrum disorders. Int Rev Psychiatry. 2018 Feb;30(1):25-39. doi: 10.1080/09540261.2018.1432574. Epub 2018 Mar 14. PMID 29537331
- [Background] Morel A, Peyroux E, Leleu A, Favre E, Franck N, Demily C. Overview of Social Cognitive Dysfunctions in Rare Developmental Syndromes With Psychiatric Phenotype. Front Pediatr. 2018 May 3;6:102. doi: 10.3389/fped.2018.00102. eCollection 2018. PMID 29774207
- [Background] Richards C, Jones C, Groves L, Moss J, Oliver C. Prevalence of autism spectrum disorder phenomenology in genetic disorders: a systematic review and meta-analysis. Lancet Psychiatry. 2015 Oct;2(10):909-16. doi: 10.1016/S2215-0366(15)00376-4. Epub 2015 Sep 1. PMID 26341300
- [Background] Webster-Stratton C, McCoy KP. Bringing The Incredible Years(R) Programs to Scale. New Dir Child Adolesc Dev. 2015 Fall;2015(149):81-95. doi: 10.1002/cad.20115. PMID 26375193
- [Background] Williams ME, Hastings RP, Hutchings J. The Incredible Years Autism Spectrum and Language Delays Parent Program: A Pragmatic, Feasibility Randomized Controlled Trial. Autism Res. 2020 Jun;13(6):1011-1022. doi: 10.1002/aur.2265. Epub 2020 Jan 21. PMID 31961490
- [Derived] Serrano M, Elias M, Llorens M, Bolasell M, Vall-Roque H, Villalta L. Early treatment for children with mental health problems and genetic conditions through a parenting intervention (The GAP): study protocol for a pragmatic randomized controlled trial. Trials. 2024 Jul 20;25(1):496. doi: 10.1186/s13063-024-08278-4. PMID 39033111

DOCUMENTS (1):
  • Study Protocol (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT06125093/Prot_000.pdf